CLINICAL TRIAL: NCT01516372
Title: A Randomized, Double-blind, Single Dose Crossover Study to Assess the Effect of Gabapentin Enacarbil on Cardiac Conduction as Compared With Placebo and Moxifloxacin in Healthy Volunteers
Brief Title: A Study to Evaluate the Effect of Gabapentin on Cardiac Repolarization in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 114112
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Restless Legs Syndrome
Keywords: GEn, moxifloxacin, cardiac repolarisation, QT/QTc
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Holliday Junction Resolvases; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment 1 (Experimental): Healthy Volunteers will receive Treatments ABDC
  Interventions: Drug: GEn 1200mg; Drug: Moxifloxacin Placebo
- Treatment 2 (Experimental): Healthy Volunteers will receive Treatments BCAD
  Interventions: Drug: Gen 6000 mg; Drug: Moxifloxacin Placebo
- Treatment 3 (Experimental): Healthy Volunteers will receive Treatments CDBA
  Interventions: Drug: GEn Placebo
- Treatment 4 (Experimental): Healthy Volunteers will receive Treatments DACB
  Interventions: Drug: GEn Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: GEn 1200mg — 1200 mg of Gen administered as a single dose
  Other Names: gen1200
  Arms: Treatment 1
Drug: Gen 6000 mg — 6000 mg of Gen administered as a single dose
  Other Names: gen6000
  Arms: Treatment 2
Drug: GEn Placebo — Placebo to match GEn Tablets
  Arms: Treatment 3; Treatment 4
Drug: Moxifloxacin Placebo — Placebo to match Moxifloxacin
  Arms: Treatment 1; Treatment 2
Drug: Moxifloxacin — 400 mg Moxifloxacin administered as a single dose
  Other Names: moxifloxacin 400
  Arms: Treatment 4

SUMMARY:
This will be a randomized, double-blind, placebo- controlled cross-over study to investigate the effect of GEn on cardiac repolarisation parameters compared with placebo and a positive control, moxifloxacin. Approximately 52 subjects will be recruited to the study and will take part in four dosing sessions. Subjects will receive, in a randomized order, a single dose of 1200 mg GEn, 6000 mg GEn (supratherapeutic dose), 400 mg moxifloxacin (positive control) and placebo. Twelve lead continuous ECG monitoring will be conducted from pre-dose to approximately 24 hours after dosing on Day 1 of each study session. The primary comparison of interest will be the mean change from baseline in the time-matched differences in QTcF between each GEn treatment and placebo.

DETAILED DESCRIPTION:
This is a 4-period, randomized, active-and placebo-controlled, double-dummy, double-blind cross-over study to evaluate the effect of single doses of GEn on cardiac conduction parameters in healthy subjects.

Screening will occur within approximately 28 days of the first scheduled dose of study medication. Each subject will participate in 4 dosing sessions at least one week apart. Prior to dosing in each period, the investigator will review the scheduled assessments to confirm the subject's suitability for the study including review of study entry criteria and lifestyle restrictions.

All subjects will receive single doses of GEn 1200 mg, GEn 6000 mg, moxifloxacin 400 mg and placebo in a randomized sequence.

Dosing with moxifloxacin will be in the fasted state and GEn will be administered following a standard meal. A double dummy approach will be used to maintain blinding. Thus, on each dosing day, moxifloxacin or moxifloxacin placebo will be administered in the fasted state in the morning and GEn or matched placebo will be administered 2 hours later after a standard meal.

During each treatment period, subjects will report to the clinical research unit the day before dosing (Day 1) and will remain until completion of the last assessment on Day 2. Twelve-lead ECGs including continuous Holter monitoring, clinical laboratory safety tests, vital sign measurements, physical examinations, adverse event reports, and pharmacokinetic samples will be collected throughout the study.

In each study period, cardiac conduction will be measured using a 24-hour continuous 12-lead Holter monitor from the morning of Day 1 until the morning of Day 2. Extraction of the Holter monitor data in triplicate for analysis will begin on Day 1 at timepoints indicated in the Time and Events Table (Section 4.7). These timepoints were selected to cover the Cmax of both moxifloxacin and GEn. If no clinically significant abnormalities are noted, subjects will be discharged from the clinical research unit after the completion of all assessments on Day 2 in each period. A minimum 7-day washout period will separate each treatment period. A follow-up visit will be conducted approximately 7 to 14 days after administration of the last dose of study medication in treatment period 4

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Male or female between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and estradiol less than 40 pg/ml (less than 147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method; Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit is completed.

Body weight greater than and equal to 50 kg and BMI within the range 19 - 30 kg/m2 (inclusive)

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Creatinine clearance (CrCl) greater than and equal to 80 mL/min. CrCl is estimated using the equation of Cockcroft and Gault. See study procedure manual for details on creatinine clearance calculations.
* AST, ALT, alkaline phosphatase and bilirubin less than and equal to 1.5xULN (isolated bilirubin greater than and equal to 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* Has cardiac conduction abnormalities on the screening 12-lead ECG denoted by any of the following: QTcB or QTcF interval greater than 450 msec; PR interval greater than 200 msec or less than and equal to 110 msec; Evidence of second- or third- degree atrioventricular block (AVB); Pathological Q-waves (defined as Q-wave greater than 40 msec or depth greater than 0.4- 0.5mV); Evidence of ventricular pre-excitation; Electrocardiographic evidence of complete left bundle branch block (LBBB), right bundle branch block (RBBB), incomplete LBBB; Intraventricular conduction delay with QRS duration greater than 120 msec
* The subject has a screening heart rate less than 50 or greater than 100 bpm or a systolic blood pressure greater than 140 or less than 100 mmHg or a diastolic blood pressure greater than 90 or ;ess than 60 mmHg in the semisupine position
* Subjects with a personal or family history of QTc prolongation, symptomatic cardiac arrhythmias or cardiac arrest
* Serum calcium, magnesium or potassium levels outside the reference range
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 14 drinks/week for men or greater than 7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Hormone replacement therapy and contraceptive medication will be allowed in this study.
* History of sensitivity to quinolone antibiotics, gabapentin, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females or pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History of seizures other than febrile seizures as a child.
* Subjects with a creatine kinase (CK) value of greater than the upper limit of normal that is not explainable by recent strenuous exercise and the value does not return within normal range upon retest.
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months. Has history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in QTcF (QT duration corrected for heart rate by Fridericia's formula) interval at Each time point for 6000 mg GEn and Placebo measured by ECG | Day -1-Day2

SECONDARY OUTCOMES:
Change in QTcF interval at Each time point for 1200 mg GEn and Placebo measured by ECG | Day -1-Day 2
Change from baseline in QTcF interval at each time point for moxifloxacin 400 mg and placebo measured by ECG | Day -1-Day 2
Change from baseline in QTcB (QT duration corrected for heart rate by Bazett's formula), QT for GEn (1200 mg and 6000 mg) and moxifloxacin (400 mg) and placebo measured by ECG | Day -1-Day 2
Change from baseline in PR, QRS intervals, heart rate and ECG waveform morphology for GEn (1200 mg and 6000 mg) and placebo measured by ECG | Day -1-Day 2
Change from baseline in heart rate and ECG waveform morphology for moxifloxacin (400 mg) | Day -1-Day 2
Pharmacokinetic parameters for gabapentin and moxifloxacin | Day -1-Day 2
Safety parameters: AEs, vital signs, ECGs, Columbia Suicide Severity Rating Scale (C-SSRS) and clinical laboratory parameters | Day -1-Day 2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

REFERENCES:
- [Derived] Davy M, Upward J, Arumugham T, Twomey C, Chen C, Stier B. Cardiac repolarization with Gabapentin enacarbil in a randomized, double-blind, placebo- and active-controlled, crossover thorough QT/QTc study in healthy adults. Clin Ther. 2013 Dec;35(12):1964-74. doi: 10.1016/j.clinthera.2013.10.011. Epub 2013 Nov 28. PMID 24290737